CLINICAL TRIAL: NCT03372148
Title: Evaluating the Role of Pharyngeal High Resolution Manometry and Impedance (pHRMi) in the Longitudinal Evaluation of Swallow Function in Head and Neck Cancer Patients
Brief Title: Role of Pharyngeal High Resolution Manometry and Impedance in Swallow Function of Head and Neck Cancer Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study withdrawn by PI
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00129556
Record Dates: First submitted 2017-12-08; First posted 2017-12-13 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Head and Neck Cancer; Dysphagia
MeSH Terms: conditions — Head and Neck Neoplasms; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Pharyngeal High Resolution Manometry and Impedance (pHRMi) in the Longitudinal Evaluation of Swallow Function in Head and Neck Cancer Patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- pHRMi in evaluation of swallowing function (Experimental): Pharyngeal High Resolution Manometry and Impedance (pHRMi) evaluation of swallowing function at baseline, 3 months post radiation, then at 9 months
  Interventions: Diagnostic Test: pHRMi

INTERVENTIONS:
Diagnostic Test: pHRMi — Pharyngeal High Resolution Manometry and Impedance swallowing function evaluation

SUMMARY:
Examining if the use of serial pHRMi to identify biomechanical changes in the swallow function of HNC patients treated with radiotherapy.

DETAILED DESCRIPTION:
Cancers located in the upper aerodigestive tract of the head and neck (HN) region present unique management challenges due to the crucial functions in this anatomic region along with its anatomic density. As such, cancers and the actual treatment can be functionally debilitating. Of these, the ability to effectively and safely transport a swallow bolus from the oral cavity to the esophagus is particularly important. This consideration has had a major influence regarding the optimal management for head and neck cancers as both oncologically effective and function-preserving therapies are desired. Accomplishing this therapeutic goal has been elusive due to a lack of tools that effectively and longitudinally evaluate swallow function over the course of a treatment and in follow-up. Standard of care approaches including modified barium swallow studies are typically used to characterize dysphagia once a clinical event has occurred such as pneumonia. As such, clinicians surprisingly lack a clear understanding of the natural history of head and neck cancer treatment - related swallow dysphagia (HNCTD) regardless of the treatment modality. Understanding which patient has HNCTD is especially important given increasing evidence that demonstrates that late secondary aspiration contributes to non-cancer related mortality in head and neck (HN) cancer patients.

To address this problem, the investigator hypothesizes that the use of quantitative and validated approaches to measuring dysphagia will allow the investigators to better define the heterogeneity seen in patients with dysphagia to gain insights into its prevention including the mortality risk of aspiration pneumonia the investigators recently demonstrated 1. Work to date using the quantitative patient-reported outcome (PRO) instruments, the Sydney Swallow Questionnaire (SSQ) and the MD Anderson Dysphagia Inventory (MDADI) has demonstrated that a reproducible signature of swallow scores can define dysphagia in irradiated HNC patients. Pilot work to date has also demonstrated that pressure flow analysis (PFA) with artificial neural network (ANN) of pharyngeal high resolution manometry and impedance (pHRMi) studies in a heterogeneous cohort of HNC patients can significantly predict for the risk of clinical aspiration and for pneumonia. This pilot study will investigate the use of serial pHRMi to identify biomechanical changes in the swallow function of HNC patients treated with radiotherapy and secondarily evaluate how the PFA may add to the investigators current PRO-defined swallow signature.

ELIGIBILITY:
Inclusion Criteria:

1. Previously untreated head and neck cancer of any histology receiving radiation with curative oncologic intent regardless of the treatment modality.

   1. The radiation can be with or without prior surgery as part of the untreated HNC treatment plan.
   2. The radiation can include concurrent chemotherapy or without.
2. Capable of providing informed consent.

Exclusion Criteria:

1. Potential study subjects with contraindications for the HRMi procedure:

   1. Potential study subjects with altered mental status or obtundation.
   2. Potential study subjects who cannot understand or follow instructions.
   3. Potential study subjects with suspected or known obstruction precluding safe passage of the manometry catheter.
2. Potential study subjects who are unwilling or unable to be adherent to longitudinal assessment and follow-up. This will include potential study subjects who have poor performance status at the time of study enrollment evaluation.
3. Potential study subjects who have cognitive limitations / impairments that prevent a potential study subject's ability to provide self-reporting with the SSQ and the MDADI instrument.
4. Potential study subjects who have motor skill limitations that prevent a potential study subject's ability to provide self-reporting with the SSQ and MDADI instrument.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Change in swallowing function as assessed by serial pHRMi | Baseline, 3 months 9 months
  Use of serial pHRMi to identify biomechanical changes in the swallow function of HNC patients treated with radiotherapy.

SECONDARY OUTCOMES:
Change in peak flow swallow measures | 9 months
  Analyze data to develop a classifier model for swallow function.

CONTACTS AND LOCATIONS:
Overall Officials: Harry Quon, MD, Principal Investigator — SKCCC at Johns Hopkins (East Baltimore Campus)
Locations (2):
- United States (2):
  - SKCCC at Johns Hopkins (East Baltimore Campus), Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No